CLINICAL TRIAL: NCT04844177
Title: Pilot Prospective Clinical Study of Safety and Efficacy of Conditioning Regimen With Total Lymphoid Irradiation Before Allogeneic Hematopoietic Stem Cell Transplantation With TCRab/CD19 Graft Depletion in Severe Congenital Neutropenia
Brief Title: Total Lymphoid Irradiation Pre-HSCT in Severe Congenital Neutropenia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2021-02
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Severe Congenital Neutropenia; GATA2 Deficiency
MeSH Terms: conditions — Neutropenia, Severe Congenital, Autosomal Recessive 3; GATA2 Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental): Total lymphoid irradiation 4 Gy (days -7, -6) in combination with:
  * Fludarabine 150 mg/m2 (days-6, -5, -4, -3, -2)
  * Cyclophosphamide 120 mg/kg (days -5, -4, -3)
  * Thymoglogulin (Genzyme) 5 mg/kg (days -5, -4)
  * Melphalan 180 mg/m2 (day -2)
  * Rituximab 100 mg/m2 (day -1)
  * Hematopoietic stem cell graft infusion after TCRab/CD19 depletion - day 0
  Interventions: Other: conditioning with TLI

INTERVENTIONS:
Other: conditioning with TLI — Total lymphoid irradiation 4 Gy (days -7, -6) in combination with:
  * Fludarabine 150 mg/m2 (days-6, -5, -4, -3, -2)
  * Cyclophosphamide 120 mg/kg (days -5, -4, -3)
  * Thymoglogulin (Genzyme) 5 mg/kg (days -5, -4)
  * Melphalan 180 mg/m2 (day -2)
  * Rituximab 100 mg/m2 (day -1)
  * Hematopoietic stem cell graft infusion after TCRab/CD19 depletion - day 0

SUMMARY:
Severe congenital neutropenia (SCN) is a group of primary immunodeficiencies caused by distinct gene mutations and characterized by neutrophil maturation impairment, which leads to neutropenia, predisposition to severe bacterial and fungal infections, and myeloid malignancies. Granulocyte-colony stimulation factor is used for pathogenetic therapy, however, no adequate response is seen in some patients.

The only curative option for SCN is hematopoietic stem cell transplantation (HSCT). An indication for HSCT in SCN is: no adequate response to G-CSF therapy, or development of malignancies, or found unfavorable mutations of SCN genes, leading to poor response to G-CSF and high risk of malignant transformation.

One of the major peculiarities of HSCT in SCN is a high risk of graft failure. That was described in few studies in SCN transplantation and was also observed in our SCN HSCT cohort. We also consider the role of TCRab/CD19 graft depletion, which is routinely used in our center for GVHD prophylaxis in increased risks of graft failure.

Another problem often observed in our patients is the relatively high risks of death of infections, developed after graft failure.

Due to predominantly early HSCT graft failure development, non-sufficient immuablation is presumed as the main reason for graft failure. Because of the low level of toxicity, associated with TCRab/CD19 depletion usage, this strategy is planned to be used in the current study. To increase an immunoablative potential of conditioning regimen in SCN, total lymphoid irradiation will be studied in combination with myeloablative agents and standardly used serotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indications for HSCT in SCN: clinical diagnosis of SCN with (1) no adequate response to G-CST therapy or (2) with malignant transformation or (3) unfavorable mutations of known SCN genes
* GATA2 deficiency
* SCN patients age at HSCT 18 months - 21 years
* GATA2 deficiency patients age at HSCT more than 10 years
* Signed informed consent to participate in the study
* Presence of HLA-matched unrelated or HLA-mismatched related donor

Exclusion Criteria:

* Presence of HLA matched related donor in absence of pathologic SCN gene mutation
* Inability to perform TCRab/CD19 graft depletion
* Contraindications for HSCT due to patients somatic condition

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-14 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years post HSCT
event free survival | 2 years post HSCT
  events - death, graft failure, secondary malignancy, relapse of malignancy

SECONDARY OUTCOMES:
Cumulative incidence of transplant related mortality | 2 years post HSCT
Cumulative incidence of graft failure | 2 years post HSCT
  non-engraftment, secondary graft rejection, severe non-reversible bone marrow failure
Cumulative incidence of graft versus host disease | 2 years post HSCT
number of patients with donor chimerism | 2 years post HSCT
Incidence of secondary malignancies | 2 years post HSCT
  number of patients
Cumulative incidence of engraftment | 100 days post HSCT
Incidence of early severe organ toxicity | 100 days post HSCT
  number of patients
cumulative incidence of infectious complications | 1 year after HSCT
  infectious complication - CMV, EVB, ADV reactivation

CONTACTS AND LOCATIONS:
Locations (1):
- HSCT department, Moscow, Russia